CLINICAL TRIAL: NCT06587711
Title: Application of Cheek Acupuncture in Vaginal Tightening Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Chunmei Chen, Attending physician, The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PlasticSurgeryHPecking
Record Dates: First submitted 2024-08-31; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pain Vulva
Keywords: Acupuncture; Analgesia; Vaginal tighting surgery
MeSH Terms: conditions — Vulvodynia; Agnosia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cheek acupuncture treatmnet (Experimental): Patients in the experimental group are treated with cheek acupuncture.
  Interventions: Procedure: acupuncture treatment
- sham acupuncture treatment (Sham Comparator): Patients in the control group are treated with sham acupuncture.
  Interventions: Procedure: acupuncture treatment

INTERVENTIONS:
Procedure: acupuncture treatment — Patients in experimental group received acupuncture at specific acupoint on the face, patients in control group received sham acupuncture at non-acupoint on the face.

SUMMARY:
A large number of studies have shown that acupuncture can reduce perioperative pain in patients. Cheek acupuncture therapy is a new acupuncture treatment, which belongs to the microneedle system, that is, acupuncture at specific acupoint on the face, which can relieve patients' pain. In this study, the efficacy and safety of cheek acupuncture in patients undergoing vaginal tightening surgery was verified by observing the consumption of opioid, intraoperative hemodynamics, dosage of oral remedial analgesics, postoperative quality of recovery, patient satisfaction, incidence of side effects, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years, undergoing vaginal tightening surgery
* American Society of Anesthesiologists (ASA) physical status I to II
* Voluntary participation and signed an informed consent form

Exclusion Criteria:

* Acute and/or chronic pain before surgery
* History of congenital heart disease, arrhythmia, or hypertension
* History of severe mental or neurological diseases, drug or psychotropic drug abuse
* Cognitive dysfunction or inability to communicate.
* The acupuncture acupoints are infected
* Coagulation disorders
* Patients with mandibular or zygomatic bone osteotomy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Intraoperative opioid consumption | End of surgery
  Intraoperative remifentanil dosage Intraoperative remifentanil dosage Intraoperative remifentanil consumption

SECONDARY OUTCOMES:
Patient intravenous controlled analgesia (PCIA) pump consumption | 24 hours after surgery
  PCIA pump consumption in 24 hours after surgery
the rest numerical rating scale (NRS) scores | 24 hours after surgery, 48 hours after surgery
  0~11，a higher score means a better outcome
the coughing numerical rating scale (NRS) scores | 24 hours after surgery, 48 hours after surgery
  0~11，a higher score means a better outcome
15-item quality of recovery (QoR-15) | 1 day after surgery, 2 day after surgery
  0~150, a higher score means a better outcome
Athens Insomnia Scale (AIS) | 24 hours after surgery, 48 hours after surgery
  0~24, a lower score means a better outcome
Hospital Anxiety and Depression Scale（HADS） | 24 hours after surgery, 48 hours after surgery
  HADS(A) and HADS(D), 0~21, respectively, a lower score means a better outcome
Patient satisfaction | 48 hours after surgery
  patient satisfaction on a Likert scale (1~5,a higher score means a better satisfaction)
Systolic blood pressure (SBP) | Enter the operating room,15 minutes after anesthesia administration, surgery onset, 1 hour of surgery, end of surgery
  Intraoperative hemodynamics
Diastolic blood pressure (DBP) | Enter the operating room,15 minutes after anesthesia administration, surgery onset, 1 hour of surgery, end of surgery
  Intraoperative hemodynamics
Mean blood pressure (MBP) | Enter the operating room,15 minutes after anesthesia administration, surgery onset, 1 hour of surgery, end of surgery
  Intraoperative hemodynamics
Heart rate (HR) | Enter the operating room,15 minutes after anesthesia administration, surgery onset, 1 hour of surgery, end of surgery
  Intraoperative hemodynamics
Opioid-related side effects | 0~48 hours after surgery
  postoperative nausea and vomiting (PONV), dizziness, headache, pruritus, and respiratory depression
Acupuncture-related side effects | 0~48 hours after surgery
  hematoma，infection
Intraoperative dexmedetomidine consumption | End of surgery
Intraoperative midazolam consumption | End of surgery
Respiratory rates (RR) | Enter the operating room,15 minutes after anesthesia administration, surgery onset, 1 hour of surgery, end of surgery
the partial pressure of end-tidal carbon dioxide (PetCO2) | Enter the operating room,15 minutes after anesthesia administration, surgery onset, 1 hour of surgery, end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yang Dong, doctorate, Study Chair — Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China